CLINICAL TRIAL: NCT04864938
Title: Recovery After Critical Covid-19 Infection
Acronym: RECOVID
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Helsinki (Other)
Collaborators: Uppsala University (Other); Göteborg University (Other)
Responsible Party: Principal Investigator, Johanna Hastbacka, Adjunct professor, University of Helsinki
Other Study IDs: HUS/1949/2020
Record Dates: First submitted 2021-02-09; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Covid-19
Keywords: intensive care unit; cognitive function; delirium; post-traumatic stress
MeSH Terms: conditions — COVID-19; Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — After separate informed consent whole blood specimens have been collected for ApoE allele analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients: ICU treated covid-19 patients: Neuropsychologic testing Respiratory function testing, chest x-ray and 6 minute walk test MRI of the brain and heart Laboratory tests Olfactory function tests Neuropsychology questionnaires
- Control group 1, covid-19 patients treated in the regular wards: As above, without 6 minute walk test or routine chest x-ray
- Control group 2, persons with covid-19 without hospitalization: As above, but without respiratory testing
- Control group 3, non-covid controls: As control group 2

SUMMARY:
The study focuses on the recovery of respiratory, cardiovascular and neurological/neuropsychological recovery after intensive care treatment for covid-19. The results will be compared with those obtained from patients treated in the regular wards for covid-19, persons with home treated covid-19 and non-covid controls.

DETAILED DESCRIPTION:
Eligible patients who have been treated in the intensive care units of Helsinki University Hospital are invited to participate. Controls are recruited from follow-up clinics, and with announcements in media and websites.

The participants receive an invitation to a follow-up clinic where their experiences from the ICU treatment and recovery will be discussed. The investigators will perform neuropsychologic testing (6 months post-discharge), a telephone interview (3 months) and send written questionnaires (3, 6 and 24 months) to the participants. The participants will undergo MRI imaging of the brain and laboratory tests will be taken. The olfactory function will be tested at a follow-up clinic. Data on the patients´ respiratory function from clinical spirometry and diffusion capacity testing 3 and 6 months after discharge are collected. The patients will perform a 6 min walk test.

Data on coagulation laboratory values will be registered from acute phase and 6 months after discharge. The investigators will also analyse ApoE alleles, neurofilament light and NAD-metabolites and study their correlation with neuropsychologic findings and long term symptoms (up to 5 years after hospital discharge).

Participants will also undergo magnetic resonance imaging of the heart at 6-12 months after the hospital discharge, and laboratory samples, a symptom questionnaire and electrocardiogram are collected. Inflammatory parameters and variables associated with regulating inflammation and coagulation will be analysed.

Clinical data from the acute and post-acute phase and demographic data are collected from the patient data management systems.

The target patient number is 75 intensive care treated patients and 50 control persons in each three control group.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-100
* Positive PCR for Sars-CoV-2 (except non-covid controls, who must be negative)
* Native language Finnish or Swedish
* Informed consent to study to study participation

Exclusion Criteria:

* Age under 18
* Pregnant or lactating
* Major neurologic diagnosis (TBI, dementia, stroke, Parkinson´s disease before covid-19)
* Substantially impaired hearing or vision
* Developmental disability.
* No consent to study participation
* Contraindication to MR imaging (such as cardiac pacemaker, allergy to contrast)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are recovering from critical covid-infection and controls that are either patients recovering from a hospital regular ward treated for covid or covid that has not required hospitalisation. Non-covid controls are age and sex-matched persons (matched to ICU treated group of participants) with no covid-19 in history.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-07-25 (Estimated); Study Completion 2024-07-25 (Estimated)

PRIMARY OUTCOMES:
Cognitive function 6 months after hospital discharge | 6 months after hospital discharge
  Global score calculated from three domains: memory, executive functions and attention.Memory: WMS-III Word list delayed recall + WMS-III Logical memory delayed recall + Rey Complex Figure, delayed recall Executive: TMB (time, reversed) + Stroop interference (time, reversed) + FAB score Attention: WAIS-IV Coding + CPT (correct items) + Stroop naming (time, reversed) The global score will be compared with controls and age matched national references
Diffusion capacity 6 months after hospital discharge | 6 months after hospital discharge
  Diffusion capacity DLCO results (percentage of predicted) 6 months after ICU treatment for covid-19
Incidence of post myocarditis findings in MRI of the heart | 6-12 months after hospital discharge
  Incidence of findings in cardiac MRI indicating previous myocarditis in each group
Six minute walk test distance | 6 months after hospital discharge
  The distance in meters walked by ICU treated patients in 6 minutes in controlled test environment
Restriction in lung function tests | 6 months after hospital discharge
  Restriction in lung function parameters vital capacity and forced vital capacity (z-scores) in measured by spirometry
Cerebral microbleeds | 6 months after hospital discharge
  Number and anatomical distribution of cerebral microbleeds in MRI imaging of the brain
Plasma matrix metalloproteinases -8, -9 and TIMP-1 6 months after hospital discharge | 6 moths after hospital discharge
  Plasma matrix metalloproteinases -8, -9 and TIMP-1 levels in ng/mL 6 months after hospital discharge
Plasma neurofilament level and its correlation with global score in neuropsychological test battery | 6 months after hospital discharge
  Plasma neurofilament level and its correlation with global score in neuropsychological test battery

SECONDARY OUTCOMES:
Correlation ApoE 4 alleles with disease severity | 6 months post-covid
  Laboratory analysis of ApoE alleles and comparison of their frequencies among groups
Correlation of cerebral microbleeds with neuropsychological global score | 6 moths after hospital discharge
  Correlation of type and location of cerebral microbleeds with neuropsychological global score
Association of the incidence of cerebral microbleeds with findings in cardiac MRI | 6-12 months after hospital discharge
  Association of the incidence of cerebral microbleeds with findings in cardiac MRI
Correlation of plasma neurofilament with cerebral microbleeds | 6 months after hospital discharge
  Correlation of plasma neurofilament with cerebral microbleeds in brain MR imaging
Correlation of 6 minute walk test heart rate variables with cardiac function | 6-12 months after hospital discharge
  Correlation of heart rate in rest, exercise and 5 minutes after exercise with cardiac output measured in heart MRI
Correlation of matrix metalloproteinase 9 with diffusion capacity | 6 months after hospital discharge
  Correlation of matrix metalloproteinase 9 (ng/mL) with lung diffusion capacity z-score

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki University Hospital, Helsinki, Capital Province of Finland, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ollila H, Pihlajamaa J, Martola J, Kuusela L, Blennow K, Zetterberg H, Salmela V, Hokkanen L, Tiainen M, Hastbacka J. Brain magnetic resonance imaging findings six months after critical COVID-19: A prospective cohort study. J Crit Care. 2024 Apr;80:154502. doi: 10.1016/j.jcrc.2023.154502. Epub 2023 Dec 19. PMID 38113746
- [Derived] Halvorsen P, Hultstrom M, Hastbacka J, Larsson IM, Eklund R, Arnberg FK, Hokkanen L, Frithiof R, Wallin E, Orwelius L, Lipcsey M. Health-related quality of life after surviving intensive care for COVID-19: a prospective multicenter cohort study. Sci Rep. 2023 Oct 21;13(1):18035. doi: 10.1038/s41598-023-45346-2. PMID 37865685
- [Derived] Ollila H, Pihlaja R, Koskinen S, Tuulio-Henriksson A, Salmela V, Tiainen M, Hokkanen L, Hastbacka J. Long-term cognitive functioning is impaired in ICU-treated COVID-19 patients: a comprehensive controlled neuropsychological study. Crit Care. 2022 Jul 20;26(1):223. doi: 10.1186/s13054-022-04092-z. PMID 35858899